CLINICAL TRIAL: NCT06244433
Title: Risk Stratification of Sudden Unexpected Death in Infant Based on Biomarkers - Identification of Genetic Variants Associated With Unexpected Infant Death Syndrome
Brief Title: Identification of Genetic Variants Associated With Unexpected Infant Death Syndrome
Acronym: BIOMINRISK
Status: Recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Collaborators: AXA Assurances VIE Mutuelle (Unknown); Institut du Thorax (Unknown)
Responsible Party: Sponsor
Other Study IDs: RC23_0260
Record Dates: First submitted 2024-01-25; First posted 2024-02-06 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2024-09

CONDITIONS: Sudden Infant Death; Sudden Unexplained Infant Death
MeSH Terms: conditions — Sudden Infant Death | interventions — Whole Genome Sequencing

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — blood and DNA samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SUDI cases: Sudden unexpected death in infant (SUDI) cases registered within the French National Registry of SUDI
  Interventions: Genetic: whole genome sequencing
- Parents: Both parents of identified SUDI
  Interventions: Genetic: whole genome sequencing

INTERVENTIONS:
Genetic: whole genome sequencing — Study of all coding and non-coding sequences in the genome to identify pathogenic allelic variants

SUMMARY:
This is a multicenter genetic study aimed at identifying new genes/variants associated with sudden infant death syndrome (SIDS) based on whole-genome sequencing of family trios

DETAILED DESCRIPTION:
The present project is part of a more global project called BIOMINRISK for which 3 axes will be explored: Genetics (a project which will be detailed here), Neurobiology and Radio-anatomical.

This is a multicenter (15 centers), national, non-randomized, open-label, genetic study. Sudden unexpected death in infant (SUDI) cases will be included (i) partly retrospectively (infants already included in the national French SUDI registry) and (ii) for the other cases, prospectively at the time of care of the deceased infant by the referral center of SUDI participating in the project. The parents making up the trios will be included prospectively.

Once the Sudden infant death syndrome (SIDS) cases have been identified among all the included SUDI cases (following the results of post-mortem examinations), Whole Genome Sequencing (WGS) will be carried out on these SIDS cases and their two parents, in order to identify pathogenic allelic variants. The data generated by this sequencing will then be analyzed using a trio approach to search for de novo variants, i.e. variants present in the infant who died of SIDS and absent from the genome of both parents.

ELIGIBILITY:
Child Inclusion Criteria

* Death of a child between 0 and 2 years of age due to sudden unexpected death in infant
* Child included in the French SUDI registry with effective participation in the biocollection
* Children who also meet the inclusion criteria for the BIOMINRISK-NEUROBIO (axis 2) and BIOMINRISK-RADIO-ANAT (axis 3) studies in the overall BIOMINRISK project.

Parents Inclusion Criteria

* Biological parents of the child included in the BIOMINRISK study
* Parents who have both signed the consent form for blood collection and inclusion of their samples in the biocollection
* parents beneficiaries of a social security or similar scheme

Child Exclusion Criteria:

* Presence of a known metabolic, genetic or syndromic pathology at the time of death

Parents Exclusion Crtiteria:

* Parent under guardianship
* Presence of a known metabolic, genetic or syndromic pathology

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The population included will consist of infants who died in the context of SUDI and both their parents. These cases of SUDI will come from the French SUDI registry, which records all cases of SUDI occurring in children under 2 years of age throughout France via a network of referral centers for the management of SUDI.
Sampling Method: Non-Probability Sample
Enrollment: 650 (Estimated)
Dates: Start 2024-08-27 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Identification of genetic variants | up to 38 months
  Presence of de novo genetic point mutations in coding and non-coding sequences, based on analysis of family trios using a whole-genome sequencing approach

SECONDARY OUTCOMES:
Identification of heterozygous variants or CNVs (copy number variants) | up to 38 months
  Presence of composite heterozygous variants or CNVs (copy number variants) in the coding and non-coding sequences of the MSN propositus genome
Identification of new genotype - phenotype correlations | up to 38 months
  Presence of new correlations between identified genetic variants and clinical and biological characteristics identified

CONTACTS AND LOCATIONS:
Overall Officials: Fleur Lorton, Principal Investigator — Nantes University Hospital
Locations (15):
- France (15):
  - Nantes University Hospital, Nantes, Loire-Atlantique
  - CHU Amiens, Amiens
  - CHU Angers, Angers
  - CHU Besançon, Besançon
  - APHP - Hôpital Jean Verdier, Bondy
  - CHU Brest, Brest
  - APHP - Hôpital Antoine Béclère, Clamart
  - CHU Grenoble, Grenoble
  - HCL, Lyon
  - AP-HM, Marseille
  - CHU Montpellier, Montpellier
  - CHRU Nancy, Nancy
  - CHU Rouen, Rouen
  - CHU Saint Etienne, Saint-Etienne
  - CHU Toulouse, Toulouse

REFERENCES:
- [Derived] Ducloyer M, Baruteau AE, Franco P, Guyon A, Sapin V, Karakachoff M, Savall F, Schott JJ, de Pontual L, De Visme S, Ferrand L, Jarry B, Beudin D, Scherdel P, Lorton F. Identification of novel genetic, neurobiological and radio-anatomical biomarkers for risk stratification of sudden unexpected death in infancy and early childhood: the BIOMINRISK study protocol. BMJ Open. 2025 Jul 30;15(7):e101811. doi: 10.1136/bmjopen-2025-101811. PMID 40738637